CLINICAL TRIAL: NCT00194272
Title: Two-Dose Methotrexate for Ectopic Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Kurt T Barnhart, MD, MSCE, University of Pennsylvania
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 701460; RRU001
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2011-08-09 (Estimated); Status verified 2011-08

CONDITIONS: Ectopic Pregnancy
Keywords: Ectopic pregnancy; Methotrexate
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Methotrexate — Two dose methotrexate
  Other Names: Rheumatrex Dose Pack; Trexall

SUMMARY:
This study examines the safety and acceptability of a novel "two dose" regimen of methotrexate to treat ectopic pregnancy.

DETAILED DESCRIPTION:
The regimen is an attempt to create a middle ground between the 2 commonly used regimens - "single dose" and "multi dose". The "multi dose" regimen is more effective, but the "single dose" regimen is more convenient for patients and has fewer side effects.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ectopic pregnancy via

  * D&E without products of conception identified on frozen pathology or
  * VABRA without products of conception identified with pathologic evaluation or
  * Ultrasound visualization of a gestational sac in the adnexa, with definitive visualization of a yolk sac or fetal pole
* the subject is hemodynamically stable without signs of hemoperitoneum
* laparoscopy has not been performed
* the subject is able to return for frequent follow-up care
* normal renal and liver function have been documented within 2 days
* normal white blood count and platelet count have been documented as per laboratory standard
* normal chest x-ray was obtained if the subject has a history of pulmonary disease
* no history of allergy or sensitivity to methotrexate or any component of its formulation

Exclusion Criteria:

* breastfeeding
* laboratory evidence of immunodeficiency
* alcoholism or chronic liver disease
* the concomitant use of non-steroidal anti-inflammatory drugs
* blood dyscrasia such as leukopenia, thrombocytopenia, or severe anemia
* active pulmonary disease
* hepatic, renal, or hematological dysfunction
* adnexal mass > or = 3.5 cm
* presence of fetal cardiac motion
* active major psychiatric disorder such as major depression, bipolar disease, psychotic disorder, or drug addiction
* subjects unable or unwilling to comply with study procedures or illiterate

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-03; Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Prevalence of side effects | Till quantitative bhCG values fall to zero or below 5mIU/mL

SECONDARY OUTCOMES:
Efficacy of treatment of ectopic pregnancy (defined as no surgical intervention) | Till quantitative bhCG values fall to zero or below 5mIU/mL

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Southern California Women's and Children's Hospital, Los Angeles, California
  - University of Miami, Miami, Florida
  - University of Pennsylvania Reproductive Research Unit, Philadelphia, Pennsylvania